CLINICAL TRIAL: NCT06259955
Title: The Effect of Mindfulness Program on Clinical Stress, Clinical Decision Making and Personality Traits in Nursing
Brief Title: The Effect of Mindfulness Program on Clinical Stress Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatma Betül Öz, Lecturer, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GazıUnıversity-Nursıng-FBOz
Record Dates: First submitted 2024-01-24; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Stress
Keywords: clinical stress; Nursing students; clinical decision; mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The trainings were conducted in Gazi University Faculty of Health Sciences Seminar Hall and Nursing Practice Laboratory with one group on Monday and Tuesday and the other group on Wednesday and Thursday. Students could miss the eight-session program at most two times. It was planned to make up for the absent course in consultation with the instructor. 37 Students attended the training regularly.
  Interventions: Other: Mindfulness
- control group (No Intervention): Throughout the study, the control group continued its routine lecture and clinical practice program. They were called only at the end of the course for the pre-test, interim measurement and post-test on the course days.

INTERVENTIONS:
Other: Mindfulness — In the hybrid education process, the group that received their first year education online realized their first face-to-face clinical practice this year. In the fall semester, internal medicine nursing course and practice, and in the spring semester, surgical diseases nursing course and practice. These two practice areas, which have a high tendency to make medical errors, require clinical decision-making skills and increase stress levels, constitute the beginning of clinical practice. Studies show that the most stressful period for students is the second year of their education (Alzayyat & Al- Gamal, 2014; White, 2011; Coram, 2015). This is because their professional knowledge and skills are not yet fully developed and they are not sufficiently prepared to meet the demands for higher level knowledge and skills (Alzayyat & Al- Gamal, 2014; Coram, 2015). Based on the results of these studies, our study group consisted of second-year students.
  Arms: intervention group

SUMMARY:
Nurses are important members of the team in the provision of health services, which determine and help the health needs of the individual, family and society, while working towards the protection and development of health, as well as taking responsibility in therapeutic services. Nurses, who are permanent members of the professional health team, need to be trained with certain skills for effective nursing care while they are still in the education process. These skills are essential skills in practice, such as critical thinking, clinical decision making, communication, creativity, coping with stress, and problem solving. The education process consists of two parts, theoretical and practical, in order to develop these skills. Clinical practical training is the cornerstone of nursing education.

Clinical practice helps to provide effective and quality care by increasing the psycho-motor skills, analysis ability and clinical decision-making skills of the student. In studies conducted with nursing students, it is seen that clinical practices are among the most important sources of stress.

Considering the reasons for the stress they experience in practice; practice for the first time, fear of making mistakes, harming the patient, difficulty in making clinical decisions, communication with nurses, lecturers and friends, lack of information, and self-confidence problems.

It is seen in the results of studies that students who experience stress in clinical practice have difficulty in decision making, decrease in their performance and self-confidence, decrease in professional career motivation, and a high tendency to make medical mistakes. Strategies for coping with stress are important when experiencing and managing stress. There are two types of coping strategies: problem-based and emotion-based. While problem-based coping aims to change the stressful event, the aim of emotion-based coping is to suppress and manage the emotions related to the stressful event. Stress mechanism and levels do not show effective results through problem-based coping alone. Emotion-based coping processes are also important. Orientation programs, simulation trainings, and laboratory practices with nursing students focus only on the knowledge level of clinical stress.There is also a need for studies on the emotional aspect of stress in the application areas. Being able to cope with stress effectively is important for students to benefit from the theoretical and clinical education they receive in a quality manner, to create a good experience and professional identity, and to develop effective coping behaviors.

DETAILED DESCRIPTION:
It is seen that clinical use with nursing beds is at the beginning of the most important stress periods. Take a look at the reasons for the stress they experience in practice; practice for the first time, fear of offspring, harming the past, difficulty in clinical decision making, communication with administrators, faculty members and friends, lack of knowledge, and lack of self-confidence. It is seen in the results of studies that students who experience stress in the clinic have difficulty in making decisions, decrease in performance and self-confidence, decrease in career motivation, and not making clean mistakes.

White reported that high anxiety measures are at the forefront of emotional states after making a clinical decision in the workplace. After an observation made by Coram , it was decided that students' anxiety caused their self-confidence to decrease and that it would negatively affect their ability to provide clinical care necessary to provide care safely. An observation made at the University of Pittsburgh is that Observation students are more successful in reaching the clinical examination than students with high self-confidence and low stress levels. Sharpnack et al. Its actions are intended to prevent appropriate clinical decision making in maternity students because of their high anxiety.

It is important for physicians working at the forefront of patient care to make good choices and make sound clinical decisions to ensure quality care.

Nursing education gains importance in the planning of the activities of various educators in providing students with aspects of clinical management coping with stress, improving clinical decision-making skills and the consequences of productive error managers.

Developing the ability to cope with stress in nursing students provides a basis for improving their clinical decision making. Conscious planning configurations are used to structure the savings, savings and stress management management and productivity of computer science students. Awareness refers to an internal perception that is intended to help individuals concentrate on the present and their environment without being distracted by organs of the past or structures.

The Kabat-Zin approach defined existing concepts to show a focused and purposeful attention to the center without judgment. Considering the ease, ease of application, and potential positive effects of awareness interpretations, many countries seem to have done a great deal of empirical work on the procedures of formal educators.

Some evidence shows that adopting temperature configurations can significantly increase temperature ranges and reduce the stress, anxiety and storage of care students.

ELIGIBILITY:
Inclusion Criteria:

* Not having participated in a mindfulness study before
* Being a second year student
* Volunteering

Exclusion Criteria:

* Being a foreign national (due to the problem of speaking/understanding Turkish)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
clinical stress score | pre-test:23.05.2022/ intermediate-test: 2 weeks after pretest / post test: 2 weeks after intermediate test
  The Clinical Stress Questionnaire (CSQ) is a five-point Likert-type questionnaire consisting of 20 items to measure the initial degree of stress experienced by nursing students on the first day of clinical practice (Pagana, 1989). The questionnaire is organised under four dimensions consisting of threat, struggle, harm and benefit feelings. Each item is analysed on a 5-point scale. In the options, 0- not at all, 1- a little, 2- moderately, 3- very much, 4- very much. A minimum of 0 and a maximum of 80 points can be obtained from the questionnaire form. A low score reveals that the stress level is low, while a high score reveals that it is high.

SECONDARY OUTCOMES:
self-confidence and anxiety scores in clinical decision making | pre-test:23.05.2022/ intermediate-test: 2 weeks after pretest / post test: 2 weeks after intermediate test
  This scale developed by Krista A. White in 2014 assesses nursing students' anxiety and self-confidence in clinical decision making (White, 2014). The scale consists of two sections, self-confidence and anxiety, and these sections are scored within themselves. The scale consists of 27 questions in total. The lowest score that can be obtained from the two sub-dimensions of the scale is 27 and the highest score is 162. For both the self-confidence and anxiety sections of the scale, there are three sub-dimensions: "Using sources to obtain information and listening fully (13 questions)", "Using available information to identify the problem (7 questions)" and "Knowing and taking action (7 questions)".

OTHER OUTCOMES:
TEN-ITEM PERSONALITY TRAITS SCALE | pre-test:23.05.2022/ intermediate-test: 2 weeks after pretest / post test: 2 weeks after intermediate test
  It is a scale developed by Gosling et al. (2003) on 112 student and non-student participants to assess personality traits. In the scale, personality traits are expressed in 10 items. These personality traits are listed as 1. Extroverted, 2. Critical, combative, 3. Reliable, self-disciplined, 4. Anxious, easily frustrated, 5. Open to new experiences, complex, 6. Timid, quiet, 7. Sympathetic, warm, 8. Upset, inattentive, 9. Calm, emotionally stable, and 10. Traditional, uncreative. The scale is a seven-point Likert scale. Respondents are expected to read each statement and rate the statement that best describes them on a scale of 1 to 7 (1.completely agree, 2.partially disagree, 3.somewhat disagree, 4.undecided, 5.somewhat agree, 6.partially agree, 7.completely agree).
perceived stress scores | pre-test:23.05.2022/ intermediate-test: 2 weeks after pretest / post test: 2 weeks after intermediate test
  It was developed in 1983 by Cohen, Kamarck and Mermelste and Cronbach Alpha value was found to be 0.86. In this study, it was adapted into Turkish by Bilge, Öğce, Genç, and Oran (2007) and Cronbach Alpha value was found to be 0.81. The PSS consists of two sub-dimensions and eight items in total. Items 1, 2, 3, 7, 8 in the perceived stress sub-dimension and items 4, 5, 6 in the coping with perceived stress sub-dimension. Three items of the five-point Likert-type scale (0 never, 4 very often) consist of inverted statements (items 4, 5, 6) and five items consist of plain statements (items 1, 2, 3, 7, 8). A score of 0-20 is obtained from the perceived stress sub-dimension, 0-12 from the coping with stress sub-dimension and a total score of 0-32 is obtained from the scale. The scale is evaluated on total and subscale scores. High scores obtained from the perceived stress sub-dimension indicate a high level of perceived stress (Bilge et al, 2009).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Unıversity, Ankara, Çankaya, Turkey (Türkiye)